CLINICAL TRIAL: NCT00502905
Title: A Phase II Study of High-Dose Intravenous Busulfan and Fludarabine With Allogeneic Marrow and Peripheral Blood Progenitor Cell Transplantation for Acute Myeloid Leukemia and Myelodysplastic Syndromes
Brief Title: Busulfan and Fludarabine in Patients With AML and MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-011
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Busulfan; Busulfex; Myleran; Fludarabine; Fludarabine Phosphate; Fludara
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Busulfan; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Busulfan + Fludarabine (Experimental): Once a day for four days, Busulfan 130 mg/m^2 through intravenous catheter over 3 hours immediately after Fludarabine 40 mg/m^2 over 1 hour.
  Interventions: Drug: Busulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Busulfan — 130 mg/m^2 injected through the intravenous catheter over three hours, once a day, for four days, starting immediately after Fludarabine.
  Other Names: Busulfex; Myleran
Drug: Fludarabine — 40 mg/m^2 through a central venous catheter over one hour, once a day, for four days.
  Other Names: Fludarabine Phosphate; Fludara

SUMMARY:
Primary Objectives:

1. To administer multiple doses of an intravenous formulation of busulfan (Bu) at a dose adjusted to yield a blood drug level with a median daily area under the plasma concentration curve (AUC) of approximately 6,500 µMol-min. This dose will be given intravenously over three hours once daily for four (4) days, in combination with Fludarabine at a dose of 40 mg/m2 as preparation for bone marrow or peripheral stern cell transplantation in patients with acute myeloid leukemia or myelodysplastic syndromes.
2. To determine the outcome of Acute Myeloid Leukemia (AML)/myelodysplastic syndromes (MDS) patients undergoing treatment with this regimen. Data regarding engraftment, toxicity, relapse rate, long-term (disease-free) outcome, and overall survival will be collected.
3. To determine the safety profile of this regimen when utilized as preparation for allogeneic transplantation.
4. To describe the plasma pharmacokinetics of busulfan when administered intravenously in this regimen.

DETAILED DESCRIPTION:
Patients who agree to the optional pharmacology procedures #1 will initially receive a therapeutic test dose of busulfan to test the blood levels over time; this information will be used to determine the subsequent high-dose busulfan doses. Patients who do not agree to the optional pharmacology procedure will receive a fixed dose of busulfan as has previously been done for 3 years.

Patients in this study will then receive fludarabine through a central venous catheter over one hour, once a day, for four days. High-dose Busulfan will be injected through the catheter over three hours, once a day, for four days, starting immediately after fludarabine.

After two days of rest, the allogeneic bone marrow, peripheral blood stem cells or cord blood will then be given intravenously. Patients will receive the drug Granulocyte colony-stimulating factor (G-CSF - Neupogen) as an injection under the skin until their blood counts recover.

Patients will remain in the hospital for about 4-6 weeks. After discharge, patients will continue as outpatients in the hospital area until they are able to safely leave the immediate hospital area or for a minimum of 100 days after the transplant. Some patients may need to receive spinal taps with instillation of cytosine arabinoside and hydrocortisone several times over the year after transplantation. This is only for patients with a previous clinical history of leukemic involvement of the brain.

This is an investigational study. The FDA has approved the study drugs. Up to 200 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Acute leukemia past first remission, in first or subsequent relapse, in first remission (high-risk, i.e., cytogenetics other than t(8;21, inv 16, t(15;17)) or induction failures.
2. Myelodysplastic syndromes in any clinical stage, excluding only patients who have isolated stable mono-cytopenia and who are clinically stable.
3. Patient has not been administered any other systemic chemotherapeutic drug (including Mylotarg) within 21 days prior to trial enrollment (BMT Day -7 or BMT day -9). (Hydroxyurea and intrathecal chemotherapy is permitted).
4. No uncontrolled infection.
5. Patients up to age 65 will be eligible for this study.
6. ALLOGENEIC TRANSPLANTATION:

   Patients should have an acceptable related or unrelated volunteer donor available for a bone marrow peripheral blood progenitor cell or cord blood transplant. Bone marrow and peripheral blood cell donors should be matched for at least 5 of 6 HLA A, B and DR loci. Cord blood donors should be matched for at least 4 of 6 A, B and DR loci.
7. Life expectancy is not severely limited.
8. Pulmonary, cardio, renal and liver function tests normal.
9. In patients < 7 years pulmonary function will be assessed per pediatric BMT routine.
10. No evidence of chronic active hepatitis or cirrhosis.
11. HIV-negative.
12. Female patient is not pregnant
13. Signed informed consent.
14. Patient admitted on Sunday, or Monday to allow for pharmacokinetic directed therapy.

Exclusion Criteria:

1) Not fulfilling eligibility criteria above.

Max Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 12, 2001 through July 14, 2005. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 200 participants enrolled, four participants were excluded from the trial and did not receive treatment.
Groups:
- Busulfan + Fludarabine: Busulfan 130 mg/m^2 + Fludarabine 40 mg/m^2 given daily for four days
Period: Overall Study
Arm/Group | Busulfan + Fludarabine
Started | 196
Completed | 196
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Busulfan + Fludarabine
Number analyzed (Participants) | 196
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 103
Region of Enrollment [Number; unit: participants]
  United States | 196

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Engraftment
Description: Successful Engraftment defined as first of 3 consecutive days with Absolute neutrophil count (ANC) equal to or more than 0.5 * 10^9/L. Failure to engraft by day +30 considered primary engraftment failure. Study period one week prior to transplant through post Day 28.
Time Frame: Study period one week prior to transplant through post Day 28
Population: Analysis per protocol.
Measure: Number; unit: participants
Arm/Group | Busulfan + Fludarabine
Number analyzed (Participants) | 196
participants | 192

ADVERSE EVENTS:
Time Frame: 7 years and 7 months
Arm/Group | Busulfan + Fludarabine
Serious Adverse Events (participants affected / at risk) | 68/196
Other Adverse Events (participants affected / at risk) | 50/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan + Fludarabine (N=196)
Pericarditis (Cardiac disorders) | 1 (1)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhagic Cystitis (Renal and urinary disorders) | 7 (7)
Bell's Palsy (Nervous system disorders) | 1 (1)
Altered Mental Status (Nervous system disorders) | 4 (4)
Graft vs Host Disease (General disorders) | 15 (15)
Fever (General disorders) | 3 (3)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Plasmapheresis (General disorders) | 1 (1)
Infection (Immune system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Cardiac Failure (Cardiac disorders) | 1 (1)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 2 (2)
Death due to Relapse (General disorders) | 2 (2)
Deep Vein Thrombosis (Cardiac disorders) | 1 (1)
Elevated serum glutamic oxaloacetic transaminase (SGOT) (Hepatobiliary disorders) | 2 (2)
Ascites (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 3 (3)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemolytic Uremic Syndrome (Blood and lymphatic system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Graft Failure (General disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystectomy (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan + Fludarabine (N=196)
Allergy (Immune system disorders) | 1 (1)
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 2 (2)
Thrombosis/Thrombus (Vascular disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis/Stomatitis (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Vaginitis (Reproductive system and breast disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 2 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 3 (3)
Increased Alanine transaminase (ALT) (Hepatobiliary disorders) | 5 (5)
Veno-Occlusive Disease (Hepatobiliary disorders) | 2 (2)
Infection (Infections and infestations) | 11 (11)
Altered Mental Status (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No